CLINICAL TRIAL: NCT02243020
Title: Study MT-St-02 - Stroke - A Randomized Pilot Study Assessing Vagus Nerve Stimulation (VNS) During Rehabilitation for Improved Upper Limb Motor Function After Stroke (MicroTransponder's Vivistim System)
Brief Title: VNS During Rehabilitation for Improved Upper Limb Motor Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroTransponder Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-St-02
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Upper Limb Deficits
MeSH Terms: conditions — Stroke | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vagus Nerve Stimulation (VNS) + Rehabilitation (1) (Experimental): This group receives vagus nerve stimulation during rehabilitation. VNS and rehabilitation are the interventions.
  Interventions: Device: Vagus Nerve Stimulation (VNS)
- Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator (Active Comparator): This group receives rehabilitation and VNS, but the VNS is different than given in the other group (rehabilitation is the only true intervention in this group). It may not be as effective as the other group's settings. Both groups receive the same amount of rehabilitation.
  Interventions: Device: Vagus Nerve Stimulation (VNS)

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS)
  Other Names: VNS

SUMMARY:
The primary study objectives are to assess the safety and feasibility of the therapy, including the surgical intervention and stimulation, as well as to provide information on the appropriateness of the study test measures (assessments) and to provide a basis for sample size calculations for a larger, pivotal study.

ELIGIBILITY:
Inclusion Criteria:

1. History of ischemic stroke that occurred at least 4 months prior to enrollment, but not more than 24 months prior
2. Age >30 years and <80 years
3. Right or left sided weakness of upper extremity
4. UEFM score within designated range.
5. At least 10 degrees of wrist extension, 10° of thumb abduction/extension, and at least 10° of extension in at least 2 additional digits

Exclusion Criteria:

1. History of hemorrhagic stroke
2. Any deficits in language or cognitive functioning that hinders participation, for example, (aphasia) or unable to follow 2 step commands.
3. Significant sensory loss.
4. Presence of ongoing dysphagia or aspiration difficulties.
5. Active major neurological or psychiatric diagnosis that would likely interfere with study protocol including prior history of brain lesions (including dementia, etc.), and current alcohol abuse, drug abuse, or epilepsy.
6. Subject receiving any therapy (medication or otherwise) at study entry that would interfere with VNS (e.g. drugs that interfere with neurotransmitter mechanisms). Additionally, no psychoactive medications - including nicotine - may be used during the acute study.
7. Prior injury to vagus nerve - either bilateral or unilateral (e.g., injury during carotid endarterectomy)
8. Severe depression
9. Not considered candidate for a device implant surgery (history of adverse reactions to anesthetics, poor surgical candidate in surgeon's opinion, etc.)
10. Any other implanted device such as a pacemaker or other neurostimulator; any other investigational device or drug
11. Medical or mental instability (diagnosis of personality disorder, psychosis, or substance abuse)
12. Pregnant or plan on becoming pregnant or breastfeeding during the study period
13. Currently require, or likely to require, diathermy during the study duration
14. Any health problem requiring surveillance with MRI imaging
15. Active rehabilitation within 4-weeks prior to therapy
16. Botox injections or any other non-study active rehabilitation of the upper extremity 4-weeks prior to and during therapy
17. Severe spasticity of the upper limb

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patty Smith, Ph.D., Principal Investigator — UT Southwestern
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - UT Southwestern, Dallas, Texas
  - UT Houston, Houston, Texas

REFERENCES:
- [Result] Kimberley TJ, Pierce D, Prudente CN, Francisco GE, Yozbatiran N, Smith P, Tarver B, Engineer ND, Alexander Dickie D, Kline DK, Wigginton JG, Cramer SC, Dawson J. Vagus Nerve Stimulation Paired With Upper Limb Rehabilitation After Chronic Stroke. Stroke. 2018 Nov;49(11):2789-2792. doi: 10.1161/STROKEAHA.118.022279. PMID 30355189
- [Result] Kimberley TJ, Prudente CN, Engineer ND, Pierce D, Tarver B, Cramer SC, Dickie DA, Dawson J. Study protocol for a pivotal randomised study assessing vagus nerve stimulation during rehabilitation for improved upper limb motor function after stroke. Eur Stroke J. 2019 Dec;4(4):363-377. doi: 10.1177/2396987319855306. Epub 2019 Jun 17. PMID 31903435
- [Result] Dickie DA, Kimberley TJ, Pierce D, Engineer N, Tarver WB, Dawson J. An Exploratory Study of Predictors of Response to Vagus Nerve Stimulation Paired with Upper-Limb Rehabilitation After Ischemic Stroke. Sci Rep. 2019 Nov 4;9(1):15902. doi: 10.1038/s41598-019-52092-x. PMID 31685853
- [Derived] Dawson J, Engineer ND, Prudente CN, Pierce D, Francisco G, Yozbatiran N, Tarver WB, Casavant R, Kline DK, Cramer SC, Van de Winckel A, Kimberley TJ. Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Stroke: One-Year Follow-up. Neurorehabil Neural Repair. 2020 Jul;34(7):609-615. doi: 10.1177/1545968320924361. Epub 2020 Jun 1. PMID 32476617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from January 2016 through August 2017 at 3 US and 1 UK sites.
Groups:
- Vagus Nerve Stimulation (VNS) + Rehabilitation (1): This group receives vagus nerve stimulation during rehabilitation. VNS and rehabilitation are the interventions.
  Vagus Nerve Stimulation (VNS)
- Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator: This group receives rehabilitation and VNS, but the VNS is different than given in the other group (rehabilitation is the only true intervention in this group). It may not be as effective as the other group's settings. Both groups receive the same amount of rehabilitation.
  Vagus Nerve Stimulation (VNS)
Period: Overall Study
Arm/Group | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: NOTE: An additional 5 subjects discontinued prior to group assignment. Three (3) discontinued due to investigator exclusion (poor surgical candidate) and two (2) self excluded (time commitment and surgical concerns). This info is as designated by the protocol and FDA device guidelines (subjects consented but were not implanted with the device).
Groups:
- Total: Total of all reporting groups
Arm/Group | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (7.4) | 60.0 (13.5) | 59.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9
  United Kingdom | 4 | 4 | 8
Time Since Stroke [Mean (Standard Deviation); unit: years] | 1.5 (.7) | 1.5 (.3) | 1.5 (.5)
Baseline Upper Extremity Fugl-Meyer (UEFM) [Mean (Standard Deviation); unit: units on a scale] | 29.5 (6.4) | 36.4 (9.4) | 33.2 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Fugl-Meyer (UEFM)
Description: Measurement of impairment, minimum value 0, maximum value 66, higher score means a better outcome. Subscales are summed.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator
Number analyzed (Participants) | 8 | 9
units on a scale | 7.6 (4.8) | 5.3 (3.2)

2. Secondary Outcome: Change in Wolf Motor Function Test Functional Assessment (WMFT)
Description: Measurement of upper limb function/mobility. For Functional Assessment - minimum is 0 and maximum is 3. A higher score means a better outcome.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator
Number analyzed (Participants) | 8 | 9
units on a scale | 0.25 (0.24) | .13 (.17)

ADVERSE EVENTS:
Arm/Group | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator
Serious Adverse Events (participants affected / at risk) | 0/8 | 3/9
Other Adverse Events (participants affected / at risk) | 4/8 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) (N=8) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator (N=9)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) — Infection at surgical site that required intravenous antibiotics. The patient recovered and the system remained implanted
Shortness of Breath and Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Shortness of breath and dysphagia due to surgical intubation. Subject improved and recovered over several weeks.
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hoarseness after surgery due to nerve manipulation. Subject's voice improved over 12 months but did not recover to 100% (significant improvement but not quite to baseline) after injection and voice therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagus Nerve Stimulation (VNS) + Rehabilitation (1) (N=8) | Vagus Nerve Stim (VNS) + Rehabilitation (2) - Comparator (N=9)
Pain/Bruising from implant surgery (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) — Pain or bruising from implant surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No